CLINICAL TRIAL: NCT02469259
Title: The Effects of Oxytocin on Social Ability, Alcohol Approach Bias, and Startle Hyperreactivity in Veterans With Alcohol Use Disorder and Post Traumatic Stress Disorder
Brief Title: The Effects of Oxytocin on Startle Hyperreactivity in Patients With AUD and PTSD
Acronym: POP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Joshua Woolley, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 15-16676
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Stress Disorders, Post-Traumatic; Alcoholism
Keywords: oxytocin; PTSD; Alcohol Use Disorder; social cognition; craving; fear-potentiated startle
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Subjects will receive either 20IU or 40IU intranasal oxytocin
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Subjects will receive intranasal saline spray
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Syntocinon
  Arms: Treatment
Other: Placebo
  Arms: Placebo

SUMMARY:
This study will investigate the effects of oxytocin on alcohol-related behaviors, social abilities, and physiological startle responses in healthy individuals and patients with posttraumatic stress disorder (PTSD) and alcohol use disorder (AUD) using a randomized, placebo-controlled, dose-tiered, between-subject study design. Specifically, the investigators will determine if intranasal administration of a single dose of the pro-social neuropeptide oxytocin decreases alcohol-related approach bias and cravings, enhances social abilities, and decreases physiological hyperactivity. The investigators will also determine the optimal dose to achieve these effects and will explore psychosocial predictors of responses to oxytocin. The proposed work has the potential to yield a novel pharmacological treatment for AUD and PTSD, both leading causes of disability in the US Military for which currently available treatments are inadequate.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75 (inclusive)
2. Current DSM-V diagnosis of PTSD
3. Current (past month) DSM-V diagnosis of a moderate to severe Alcohol Use Disorder

Exclusion Criteria:

1. Current or lifetime psychotic disorders, such as schizophrenia or bipolar disorder
2. Dementia or other neuropsychiatric disorders involving cognitive deficits or active symptoms impairing their ability to complete study tasks.
3. Subjects known to have clinically significant unstable medical conditions, including but not limited to clinically significant renal disease.
4. Use of disulfiram, naltrexone, or acamprosate for alcohol use disorder in the past week.
5. Needing acute medical detoxification from alcohol based on a score of 12 or more on the Clinical Institute Withdrawal Assessment of Alcohol Scale (CIWA-AD);
6. Subjects who are legally mandated to participate in an alcohol treatment program.
7. Subjects who have had a suicide attempt in the past 6 months or suicidal ideation in the 90 days prior to enrollment.
8. Subjects with seizure disorders that require anticonvulsant medications
9. Positive urine pregnancy test, women meeting DSM-V criteria for premenstrual dysphoric disorder or with diseases likely to influence hormonal or neuroendocrine status
10. Sensitivity to preservatives (in particular E 216, E 218 and chlorobutanol hemihydrate)
11. Nasal obstruction, discharge, or bleeding
12. Taking testosterone or estrogen/progesterone supplement, or 5HT1a agonists/antagonists, as these agents can alter oxytocin levels

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Social Perception measured by score on the Reading the Eyes in the Mind Test | Participants will complete the task 60 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Alcohol Approach Bias measured by score on the Approach Avoidance Task | Participants will complete the task 65 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Startle Hyperactivity measured by heart rate change score in response to startle stimuli | Participants will complete the task 70 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Craving will measured by heart rate change score in response to a Cue-Induced Craving task | Participants will complete the task 80 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Craving will measured by skin conductance change score in response to a Cue-Induced Craving task | Participants will complete the task 80 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Theory of Mind will me measured by score on the Theory of Mind Geometric Task | Participants will complete the task 90 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Social Threat Processing will be measured by score on the Social Dot Probe Task | Participants will complete the task 100 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Social Cognition will be measured by score on the Facemorph Task. | Participants will complete the task 105 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.
Working Memory will be measured by score on the Symmetry Span Task | Participants will complete the task 120 minutes following test drug administration. This will occur 3 times during the study period, with each visit separated by at least 7 days. The total study duration will be an average of 4 weeks per subject.

CONTACTS AND LOCATIONS:
Overall Officials: Josh D Woolley, MD/PhD, Principal Investigator — University of California San Francisco, San Francisco Veterans Affairs Medical Center
Locations (1):
- San Francisco Veterans Affairs Medical Center, San Francisco, California, United States